CLINICAL TRIAL: NCT04824014
Title: Evaluation of the Diagnostic, Prognostic and Follow-up Potential of 4,16α-[16α-18F]Difluoro-11β-methoxyestradiol (4FMFES) PET Imaging for Estrogen Receptor Positive Advanced Breast Cancers
Brief Title: 4FMFES-PET Imaging of ER+ Advanced Breast Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, MD, FRCPC, Head of clinical research, CIMS, CRCHUS, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIMS-4FMFES-2021-3966
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: ER+ Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4FMFES-PET imaging at 0, 6 and 18 months (Experimental): Patients burdened with ER+ advanced breast cancers and recruited in the trial will undergo an experimental 4FMFES-PET imaging within a 4-week interval of a medically-prescribed FDG-PET. The 4FMFES-PET procedure will be repeated at 6 and 18 months following the initial scan.
  Interventions: Diagnostic Test: 4FMFES-PET

INTERVENTIONS:
Diagnostic Test: 4FMFES-PET — Intravenous 4FMFES injection, followed with PET imaging
  Other Names: 4,16α-[16α-18F]difluoro-11β-methoxyestradiol PET

SUMMARY:
Estrogen Receptor (ER) is a crucial prognostic factor and treatment target in breast cancer patients. Knowledge of its status greatly influences the choice of the optimal course of treatment. Pathological evaluations of primary tumor, axillary nodes, and metastases are the only confirmatory approach to ER status determination and are limited to known and accessible sites. However, it is known that many advanced breast cancer patients harbor diseases presenting inter-tumor or temporal ER heterogeneity, as ER expression can vary between tumor foci and can evolve during treatment and at time of recurrence, hence the need for whole-body, non-invasive assessment of ER status.

In the last decades, 16α-[18F]fluoroestradiol (FES) was developed and evaluated as an ER-targeting positron emission tomography (PET) tracer. FES correlated with ER expression, and recently was shown to be able to predict hormone therapy response. Our Center designed and evaluated 4-fluoro-11β-methoxy-16α-[18F]fluoroestradiol (4FMFES), a successor PET tracer for ER imaging. Paired comparison during a phase II clinical trial showed that 4FMFES produced images of better quality, with less overall non-specific signal than FES. It resulted in a significantly improved tumor contrast and tumor detectability using 4FMFES-PET leading to increased diagnosis confidence in early-stage breast cancer compared to FES-PET. Those results demonstrated that, as of now, 4FMFES-PET is the best imaging modality worldwide for whole-body ER status determination, but further validations are necessary to position this method as a standard and essential tool for breast cancer management. Like what was observed for FES-PET, preliminary data suggest that 4FMFES-PET combined with FDG-PET will yield very high sensibility for breast tumor detection, each method being complementary.

In continuity with previous work, we seek to expand our clinical knowledge of this high-potential diagnostic imaging through the following main objective:

Launch a phase II clinical trial to explore the full potential and benefit of 4FMFES-PET in combination with FDG-PET for advanced ER+ breast cancer patients to demonstrate it is an essential tool for cancer management.

This proposed project will focus on 3 specific aims:

1. Compare and complement 4FMFES-PET with FDG-PET and conventional imaging modalities, and evaluate how they improved prognosis and staging of ER+ advanced breast cancer patients;
2. Correlate 4FMFES/FDG uptake and staging with pathological data (histology, receptor status, grade), including distal biopsy metastases sampling;
3. Correlate 4FMFES/FDG uptake and staging with longitudinal outcomes (treatment response, progression-free survival, time-to-relapse) to determine which cohort of patient benefit most from 4FMFES.

ELIGIBILITY:
Inclusion Criteria:

* Advanced breast cancer patients, i.e. stage 3 or 4 diseases.
* Aged 18 or older at the time of breast cancer diagnosis.
* Histopathologic review confirming diagnosis of ER positive breast cancer.
* Male patients, although rare, can participate.
* Patient must have given informed consent.
* ECOG performance status 0-3.
* ER must be positive in at least 10% of tumor cells in either the core biopsy or a therapeutic surgical resection.
* Any HER2-neu status.
* Patient eligible for and willing to receive systemic treatment.

Exclusion Criteria:

* Patients who are pregnant or nursing.
* Patients unable to tolerate PET/CT for 30 minutes.
* Patients taking anti-ER hormone therapy that can pharmacologically blockade estrogen receptors (ex: Tamoxifen, Fulvestrant). Patients can undergo 4FMFES-PET if anti-ER therapy was interrupted at least 8 weeks prior imaging. Aromatase inhibitors and LHRH analogs are not expected to interfere with 4FMFES uptake and are thus permitted to be taken prior and during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of 4FMFES-PET uptake with histopathological markers, notably ER immunohistochemistry (IHC) score | 18 months
  4FMFES-PET targets Estrogen Receptors (ER) in ER+ cancers with high affinity, at least in vitro. 4FMFES-PET was already compared to the similar PET tracer FES, whose uptake is known to correlate with ER status and IHC score, and shown to have superior diagnostic properties. 4FMFES-PET will now be correlated with the ER IHC score, along with other histopathological markers.
Evaluation of progression-free survival versus 4FMFES-PET uptake threshold | 18 months
  This outcome aims to evaluate the prognostic potential of 4FMFES-PET. Kaplan-Meyer curves of progression-free-survival (PFS) will be drawn, with the studied population separated with A) a 4FMFES-PET SUVMax cut-off value of 1.5; and B) FDG-PET/4FMFES-PET tumor ratio cutoff value of 2.0, each for the lowest uptake tumor within the same patient at the initial assessment. It is expected that higher 4FMFES uptake and lower FDG/4FMFES ratio will be associated with better outcome for patients.Significant differences will be evaluated using the Log-Rank test.
Evaluation of time-to-recurrence versus 4FMFES-PET uptake threshold | 18 months
  This outcome aims to evaluate the prognostic potential of 4FMFES-PET. Kaplan-Meyer curves of time-to-recurrence (TTR) will be drawn, with the studied population separated with A) a 4FMFES-PET SUVMax cut-off value of 1.5; and B) FDG-PET/4FMFES-PET tumor ratio cutoff value of 2.0, each for the lowest uptake tumor within the same patient at the initial assessment. It is expected that higher 4FMFES uptake and lower FDG/4FMFES ratio will be associated with better outcome for patients.Significant differences will be evaluated using the Log-Rank test.
Correlation of treatment response with reduction of 4FMFES-PET uptake and number of assessable lesions at 6 and 18 months after the initial assessment | 18 months
  All patients on the study will be followed longitudinally with clinical questionnaire and examination as of their treating oncologist. Clinical information on treatment details, first progression and site of progression will be recorded on a follow-up form at each visit for at least 3 years. All stage 3 breast cancer patients with a breast in place will undergo annual mammograms with or without breast ultrasound as of current standard practice.
  Patients receiving chemo-, radio and/or hormone therapy will be longitudinally followed-up using 4FMFES-PET and FDG-PET at 6 months and 18 months following the initial scan. Imaging at shorter intervals could also be done if deemed necessary. Tracer uptake, number and size of lesions will be documented at each imaging.
  If it occurs, case of death will be sought from hospital or community medical records.
Complementarity analysis of FDG-PET with 4FMFES-PET | 36 months
  4FMFES-PET will be scheduled within two weeks of a clinically prescribed FDG-PET to allow 4FMFES to FDG comparison.
  Uptake (SUV: Standardized Uptake Value) and contrast (tumor SUVMax / background SUVMean ratio) will be measured and compiled for each lesion. Detection of each lesion will be determined by the contrast value: 1) higher or equal to 3 = positive; 2) between 1.5 and 3 = ubiquitous; 3) under 1.5 = negative. A study will be considered as 4FMFES-negative if 4FMFES-PET does not display any focal uptake other than normal physiological biodistribution, and the same will be done for FDG-PET. Unsuspected lesion visible on 4FMFES-PET or FDG-PET will be investigated by biopsy when possible to prove the lesion's histopathology. Follow-up images will be compared with the initial FDG and 4FMFES-PET scans for each patient, and both the total number of visible tumors and their uptake will be compared between each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Eric E Turcotte, MD, Principal Investigator — Université de Sherbrooke, Centre de Recherche du CHUS
Locations (1):
- Université deSherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No